CLINICAL TRIAL: NCT02847442
Title: Efficacy and Safety of Opicapone in Clinical Practice in Parkinson's Disease Patients With Wearing-off Motor Fluctuations
Brief Title: Efficacy and Safety of Opicapone in Clinical Practice
Acronym: OPTIPARK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-OPC-401; 2016-002391-27 (EudraCT Number)
Record Dates: First submitted 2016-07-21; First posted 2016-07-28 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Parkinson's Disease With Wearing-off Motor Fluctuations
Keywords: Ongentys
MeSH Terms: interventions — opicapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Opicapone (BIA 9-1067) 50 mg (Experimental): Total duration of trial participation and treatment: three months. All subjects will start treatment with 50 mg opicapone (OPC) once daily for a 3-month period in addition to their current treatment with levodopa/dopa decarboxylase inhibitor (L-dopa/DDCI)
  Interventions: Drug: BIA 9-1067; Drug: levodopa/dopa decarboxylase inhibitor

INTERVENTIONS:
Drug: BIA 9-1067 — Opicapone (BIA 9-1067) 50 mg hard capsules. Oral administration, once daily at bedtime, at least one hour before or after the last daily dose of L-dopa/DDCI.
  Other Names: Ongentys; Opicapone
Drug: levodopa/dopa decarboxylase inhibitor — OPC enhances the effects of L-dopa. Hence, it may be necessary to reduce the subject's L-dopa/DDCI dose within the first days or weeks of OPC treatment by extending the dosing intervals and/or reducing the amount of L-dopa/DDCI per dose
  Other Names: L-dopa/DDCI

SUMMARY:
The purpose of this study is to evaluate the change in subject's condition according to the Investigator's Global Assessment of Change after three months of treatment with 50 mg opicapone once daily in a heterogeneous patient population reflecting daily clinical practice.

DETAILED DESCRIPTION:
This is a prospective, open-label, uncontrolled, single-group, multi-centre trial in Parkinson's disease (PD) patients with wearing-off motor fluctuations.

At screening/baseline (Visit 1, Day 1) all subjects will start treatment with 50 mg opicapone (OPC) once daily for a 3-month period in addition to their current treatment with levodopa/dopa decarboxylase inhibitor (L-dopa/DDCI). Subjects treated with L-dopa/DDCI/entacapone before trial entry will discontinue entacapone treatment at this visit. Subjects treated with L-dopa/DDCI/tolcapone before trial entry will not be eligible, as well as those previously treated with OPC. Subjects treated with dopamine agonists will be eligible.

OPC enhances the effects of L-dopa. Hence, it may be necessary to reduce the subject's L-dopa/DDCI dose within the first days or weeks of OPC treatment by extending the dosing intervals and/or reducing the amount of L-dopa/DDCI per dose. Therefore, on Day 15 ±3 (Visit 2) the investigator will call the subject to ask for adverse events (AE, e.g. dopaminergic AEs) and if required, to reduce the L-dopa/DDCI dose. The investigator may increase or decrease the total daily L-dopa/DDCI dose according to the subject's condition throughout the trial, except at Visit 1. At the Visit 1 the L-dopa dose should not be changed.

Further visits will be performed on Day 30 ±4 (Visit 3) and on Day 90 ±4 (Visit 4). Subjects who discontinue trial participation prematurely will be asked to come to the site for an early discontinuation visit (EDV).

In addition to the scheduled visits, subjects may be asked to call or to return to the trial site, or subjects may be called by the investigator for assessment of safety data or adjustment of L-dopa/DDCI dose (unscheduled visits).

At Visit 4 (or EDV, if applicable) the investigator will arrange for the subject's subsequent PD treatment, i.e. either prescribe further OPC or switch to another treatment.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign an informed consent form.
* Male and female subjects aged 30 years or older.
* Diagnosed with idiopathic PD according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria.
* Disease severity Stages I-IV (modified Hoehn - Yahr staging) at ON.
* Treated with three to seven daily doses of L-dopa/DDCI or L-dopa/DDCI/entacapone, which can include a slow-release formulation.
* Signs of "wearing-off" phenomenon according to the 9-Symptom Wearing-off Questionnaire (WOQ-9), despite optimal anti-PD therapy (based on the investigator's judgement). The wearing-off phenomenon has to be confirmed clinically by the investigator.
* For females: Postmenopausal for at least two years or surgically sterile for at least six months before screening.

Exclusion Criteria:

* Non-idiopathic PD (atypical parkinsonism, secondary [acquired or symptomatic] parkinsonism, Parkinson-plus syndrome).
* Severe OFF periods. Patients with rare and/or short unpredictable OFF periods are eligible.
* Previous or current use of tolcapone and/or OPC.
* Treatment with monoamine oxidase inhibitors (MAO-A and MAO-B; except selegiline up to 10 mg/day in oral formulation or 1.25 mg/day in buccal absorption formulation or rasagiline up to 1 mg/day or safinamide up to 100 mg/day) within the month before screening.
* Concomitant treatment with entacapone.
* Use of any other investigational medicinal product (IMP), currently or within the three months (or within five half-lives of the IMP, whichever is longer) before screening.
* Any medical condition that might place the subject at increased risk or interfere with assessments.
* Past (within the past year) or present history of suicidal ideation or suicide attempts.
* Current or previous (within the past year) alcohol or substance abuse excluding caffeine or nicotine.
* Phaeochromocytoma, paraganglioma, or other catecholamine secreting neoplasms.
* Known hypersensitivity to the ingredients of IMP (including lactose intolerance, galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption).
* History of neuroleptic malignant syndrome (NMS) or non-traumatic rhabdomyolysis.
* Severe hepatic impairment (Child-Pugh Class C).
* For females: Breastfeeding.
* Employees of the investigator, trial centre, sponsor, clinical research organisation and trial consultants, when employees are directly involved in the trial or other studies under the direction of this investigator or trial centre, and their family members.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2016-11-23 (Actual); Primary Completion 2018-07-04 (Actual); Study Completion 2018-07-04 (Actual)

PRIMARY OUTCOMES:
Investigator's Global Assessment of Change | Through study completion, an average of three months

SECONDARY OUTCOMES:
Change in L-dopa total daily dose | Through study completion, an average of 3 months
percentage of subjects with change in number of daily L-dopa doses | Through study completion, an average of 3 months
percentage of subjects with change in L-dopa single dose (SD) | Through study completion, an average of 3 months
percentage of subjects with stable L-dopa regimen | Through study completion, an average of 3 months
percentage of subjects for whom OPC will be prescribed | Through study completion, an average of 3 months
percentage of subjects who stopped treatment with OPC | Through study completion, an average of 3 months
Subject's Global Assessment of Change at Visit 3 | Through study completion, an average of 3 months
Subject's Global Assessment of Change at Visit 4 | Through study completion, an average of 3 months
Absolute values in unified Parkinson's disease rating scale (UPDRS) scale | Through study completion, an average of 3 months
Change from baseline to Visit 4 in UPDRS scale | Through study completion, an average of 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Carl Gustav Carus at the TU Dresden, Neurological University Clinic, Dresden, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Schofield C, Chaudhuri KR, Carroll C, Sharma JC, Pavese N, Evans J, Foltynie T, Reichmann H, Zurowska L, Soares-da-Silva P, Lees A. Opicapone in UK clinical practice: effectiveness, safety and cost analysis in patients with Parkinson's disease. Neurodegener Dis Manag. 2022 Apr;12(2):77-91. doi: 10.2217/nmt-2021-0057. Epub 2022 Mar 21. PMID 35313124
- [Derived] Reichmann H, Lees A, Rocha JF, Magalhaes D, Soares-da-Silva P; OPTIPARK investigators. Effectiveness and safety of opicapone in Parkinson's disease patients with motor fluctuations: the OPTIPARK open-label study. Transl Neurodegener. 2020 Mar 4;9(1):9. doi: 10.1186/s40035-020-00187-1. PMID 32345378